CLINICAL TRIAL: NCT01528410
Title: ALFApump® System Versus Large Volume Paracentesis in the Treatment of Refractory Ascites. A Multicentre Randomised Controlled Study.
Brief Title: ALFApump System Versus Standard of Care in Ascites Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-AAR-005
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Refractory or Recurrent Ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Intervention Model Description: The study will be a single center, open-label trial.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALFApump removal of ascites (Experimental): Removal of ascites
  Interventions: Device: ALFApump removal of ascites
- Large volume paracentesis for removal of ascites (Active Comparator): Removal of ascites
  Interventions: Procedure: Large volume paracentesis for removal of ascites

INTERVENTIONS:
Device: ALFApump removal of ascites — Implanted ALFApump, removing produced ascites according to programmed schedule
  Other Names: ALFApump (Automated Low Flow Ascites pump)
  Arms: ALFApump removal of ascites
Procedure: Large volume paracentesis for removal of ascites — Large volume paracentesis - standard of care, removing ascites according to patient need
  Other Names: Extraction of fluid from the abdominal cavity
  Arms: Large volume paracentesis for removal of ascites

SUMMARY:
This is a multicentre, open, randomised, and controlled trial conducted in sixty (60) patients diagnosed with refractory or recurrent ascites. Patients will be randomised (enrolled) to either treatment arm A- implanted with the ALFApump System or treatment arm B-standard of care with evacuation large volume paracentesis. The main aims of the study are to determine the paracentesis free survival, defined as the time to the first large volume therapeutic paracentesis > 5 litres. The secondary aims are to assess non-inferiority of cirrhosis-related complications in the group of patients randomized to the ALFApump system group, as well as nutritional effects, resource utilisation, patient quality of life and survival non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females (determined by serum pregnancy test) ≥ 18 years of age. Women of childbearing age must be prepared to use at least 1 effective (≤ 1% failure rate) method of contraception during the course of the study
2. Cirrhosis of the liver defined by histological and/or clinical, and/or radiological criteria
3. Presenting refractory or recurrent ascites and requiring periodic large volume paracentesis (large volume defined as > 5 L to accord with teh clinical guidance of EASL, European Association for the Study of the Liver, which recommends withdrawal of 5 L should precipitate administration of albumin).
4. Capable of giving written informed consent, willing to comply with study procedures and ability to operate the device

Exclusion Criteria:

1. Gastrointestinal haemorrhage over the last 7 days
2. Renal failure defined as serum creatinine higher than or equal to 2 mg/dl
3. Severe coagulopathy defined as prothrombin time greater than 40% more than upper limit of Normal (as determined locally).
4. Platelet count of less than 40000 /uL unless platelet therapy is given at the time of surgery
5. Clinical Evidence of recurring bacterial peritonitis, defined as 2 or more episodes over the last 6 months or a single episode within the last 2 weeks.
6. Clinical evidence of recurring urinary infections, defined as 2 or more episodes over the last 6 months or a single episode within the last 2 weeks.
7. Clinical evidence of loculated ascites.
8. Advanced hepatocarcinoma, defined as one which exceeds Milan criteria.
9. Obstructive uropathy, residual urinary volume exceeding 100 ml, or any bladder anomaly which might contraindicate implantation of the device.
10. Concurrently implanted with any other Active Implantable Medical Device, including, but not limited to, cardiac pacemaker or cardioverter defibrillator.
11. Pregnant females or females anticipating pregnancy during study period
12. Patients currently enrolled in another interventional clinical study
13. Other concomitant disease or condition likely to significantly decrease life expectancy or present anaesthetic risk (e.g., moderate to severe congestive heart failure)
14. Known presence of human immunodeficiency virus (HIV)
15. Immuno-modulatory treatment (including azothioprine, methotrexate, anti-TNF therapies) used within last 4 months
16. Known or suspected hepatic or extra hepatic malignancy, unless adequately treated or in complete remission for ≥ 3 years
17. BMI > 40 presenting a risk for surgery and tunneled lines
18. Patients with contraindications for general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-08-17 (Actual); Primary Completion 2016-09-21 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
Paracentesis free survival | 6 months
  Paracentesis-free survival, defined as time to first large volume therapeutic paracentesis > 5 litres

SECONDARY OUTCOMES:
Non-inferiority of cirrhosis related complication in the patient group treated with the ALFApump system | 6 months
  Cirrhosis-related complications
Quality of Life | 6 months
Body weight | 6 months
Nutritional profile | 6 months
Resource utilisation | 6 months
Survival | 6 months
Assess the need for repeat evacuation paracentesis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Jalan, Professor, Principal Investigator — UCL Institute of Hepatology, Royal Free Hospital, London
Locations (7):
- Vienna General Hospital and Medical School, AKH, Vienna, Austria
- France (2):
  - Hopital Beaujon, Clichy, Paris
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Azienda Ospedaliera di Padova, Padua, Italy
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- United Kingdom (2):
  - Bristol Royal Infirmary, Bristol
  - Royal Free Hospital, London

REFERENCES:
- [Derived] Stepanova M, Nader F, Bureau C, Adebayo D, Elkrief L, Valla D, Peck-Radosavljevic M, McCune A, Vargas V, Simon-Talero M, Cordoba J, Angeli P, Rossi S, MacDonald S, Capel J, Jalan R, Younossi ZM. Patients with refractory ascites treated with alfapump(R) system have better health-related quality of life as compared to those treated with large volume paracentesis: the results of a multicenter randomized controlled study. Qual Life Res. 2018 Jun;27(6):1513-1520. doi: 10.1007/s11136-018-1813-8. Epub 2018 Feb 19. PMID 29460201
- [Derived] Bureau C, Adebayo D, Chalret de Rieu M, Elkrief L, Valla D, Peck-Radosavljevic M, McCune A, Vargas V, Simon-Talero M, Cordoba J, Angeli P, Rosi S, MacDonald S, Malago M, Stepanova M, Younossi ZM, Trepte C, Watson R, Borisenko O, Sun S, Inhaber N, Jalan R. Alfapump(R) system vs. large volume paracentesis for refractory ascites: A multicenter randomized controlled study. J Hepatol. 2017 Nov;67(5):940-949. doi: 10.1016/j.jhep.2017.06.010. Epub 2017 Jun 21. PMID 28645737